CLINICAL TRIAL: NCT03791853
Title: Achieving Rapid Diagnosis During Breast Cancer Surgery Using Light-CT (High-resolution Full-field Optical Coherence Tomography and Dynamic Cell Imaging)
Brief Title: Light-CT in the Diagnosis of Breast Tumor and Lymph Node
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LightCT-PKUPH
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Optical Coherence Tomogram; Sentinel lymph node; Dynamic cell imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Light-CT: All specimens are detected using Light-CT
  Interventions: Diagnostic Test: Light-CT

INTERVENTIONS:
Diagnostic Test: Light-CT — Fresh specimen is trimmed into a block with a size not larger than 2.5 cm (Typically not larger than 1.5 cm). Prepared specimen is submitted to Light-CT tests. FF-OCT images are obtained to depict the structure information and DCI images are generated to collect the dynamic information of the cell and tissue. After the imaging detection, specimens are submitted for routine pathological diagnosis to obtain corresponding pathological images.

SUMMARY:
Intraoperative pathological diagnosis such as frozen section and imprint cytology is not routinely recommended in clinical practice because of time and accuracy concerns. Full-field optical coherence tomography (FF-OCT) is a new optical imaging technique that could generate sectioning tomogram from fresh tissue and provide close-to-pathology depiction of the morphological structure and pathological changes in minutes without conventional tissue preparation, slicing, and staining, and dynamic cell imaging (DCI) added the viability information of cells/tissue, which could be more important in cancer diagnosis. This study was to evaluate the feasibility and diagnostic value of FF-OCT and DCI in breast lesions and lymph node specimens during breast cancer surgery. We evaluated normal breast tissue, benign breast lesions, breast cancer and axillary lymph node specimens resected from patients undergoing breast surgery.

DETAILED DESCRIPTION:
Light-CT, a special-designed pathology-approximation system which is based on the lighting feature or dynamic feature of tissue and cells, is used to detect malignant cells or tissue in fresh specimens. Morphological structure and pathological changes could be captured in minutes, which implies a possible application in intraoperative diagnosis. In this study, fresh breast tissue, fat, benign breast lesions, breast cancer and axillary lymph node specimens are collected to assess the usefulness of Light-CT. During the in vitro examination, both FF-OCT and DCI images are obtained and stored. Imaging analysis would be performed in traditional imaging analysis like manner and an artificial intelligence aided approach as well.

In this study, breast and lymph node specimens would be collected and imaged both through light imaging and conventional pathological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to undergoing breast surgery/surgical lymph node staging.
* Specimen could be obtained.

Exclusion Criteria:

* Prior open biopsy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning to undergoing breast surgery and breast cancer patient planning to undergoing surgical lymph node staging are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Light-CT | One week after the release of the pathological reports.
  The true positive rate measures the proportion of positives that are correctly identified by ultrasound

SECONDARY OUTCOMES:
The lighting feature of different tissue | Through study completion, an average of 1 year
  By the comparison analysis of FF-OCT and DCI images and corresponding pathological images, lighting feature would be extracted.
Specificity of Light-CT | One week after the release of the pathological reports.
  The true negative rate measures the proportion of positives that are correctly identified by Light-CT.
Examination time | Through study completion, an average of 1 year
  The time from the specimen preparation to the completion of the examination.

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, M.D., Principal Investigator — Peking University People's Hospital
Locations (3):
- China (3):
  - Breast Center, Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing
  - Xuanwu Hospital of Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided